CLINICAL TRIAL: NCT07386808
Title: An Analysis of the Improvement of Sleep Disorders in Patients With Alzheimer's Disease After Sunlight Exposure Therapy.
Brief Title: Improvement of Sleep Disorders in Patients With Alzheimer's Disease After Sunlight Exposure Therapy.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 202511021RIND
Record Dates: First submitted 2026-01-15; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer's Disease (AD); Sleep Disorders, Circadian Rhythm
MeSH Terms: conditions — Alzheimer Disease; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Routine nursing care (Other): no additional sunlight therapy
  Interventions: Behavioral: sunlight therapy

INTERVENTIONS:
Behavioral: sunlight therapy — They were informed that sun exposure therapy could effectively improve sleep, and behavioral interventions were discussed to develop a health education plan. Telephone follow-ups were conducted on days 3, 7, 10, and 14 after enrollment to understand the sun exposure practices of the experimental group, including the duration of sun exposure, whether the light source was indoor light or sunlight, and positive encouragement was provided.

SUMMARY:
This observational study aimed to understand the effect of intervention A on sleep disorders in individuals with Alzheimer's disease receiving sunlight therapy. The primary question of the study was:

Does sunlight therapy improve sleep disorders in Alzheimer's disease?

Participants will complete a questionnaire, undergo sunlight therapy, and have their sleep patterns recorded for 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Alzheimer's disease
2. CDR: 0.5 - 1 point
3. Conscious and able to cooperate with behavioral interventions and telephone interviews
4. Complaints of sleep disturbances, including: daytime sleepiness, difficulty falling asleep, fragmented sleep, nighttime awakening, nocturnal wandering, and sunset syndrome.
5. A cohabiting family member is required as the primary caregiver, who understands and cooperates with this intervention and has signed a consent form.
6. If the patient is already taking sleeping pills, the maintenance dose will not be adjusted.

Exclusion Criteria:

1. Individuals with other brain injury conditions, such as cerebral palsy, brain tumors, traumatic brain injury, or stroke.
2. Individuals with visual impairments (assessed by comparing numbers with fingers at a distance of 30 cm upon admission).
3. Institutional residents.
4. Individuals living alone.
5. Individuals unable to cooperate with behavioral interventions and telephone interviews.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index, PSQI | on enrollment days, 7, and 14 after enrollment
  The Pittsburgh Sleep Quality Index (PSQI) assesses sleep quality. It has seven dimensions: sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, medication use, and daytime activity impairment. A higher PSQI score indicates poorer sleep quality. The total score ranges from 0 to 21, with a minimum score of 0, indicating very good sleep quality over the past month. Lower scores indicate better sleep quality, while a total score of 5 or below is generally considered to indicate fair sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided